CLINICAL TRIAL: NCT00938314
Title: A Phase IIb Prospective, Randomized, Double-blind, Placebo Controlled, Multicenter, Dose Escalation Study of NTx®-265: Human Chorionic Gonadotropin (hCG) and Epoetin Alfa (EPO) in Acute Ischemic Stroke Patients (REGENESIS-LED)
Brief Title: Study of NTx®-265: Human Chorionic Gonadotropin (hCG) and Epoetin Alfa (EPO) in Acute Ischemic Stroke Patients
Acronym: REGENESIS-LED
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: Stem Cell Therapeutics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTx®-265-CP-202-IS
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Results first posted 2011-11-09 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Chorionic Gonadotropin; Ovidrel; Epoetin Alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- NTx®-265 Low Dose (Experimental): hCG 385 µg (10,000 international unit [IU]), subcutaneously (SC), on Day 1, 3 and 5 of study participation, then EPO 4,000 IU, intravenously (IV), on Day 7, 8, and 9 of study participation
  Interventions: Drug: human chorionic gonadotropin (hCG), then epoetin alfa (EPO)
- NTx®-265 Medium Dose (Experimental): hCG 385 µg (10,000 IU), SC, on Day 1, 3 and 5 of study participation, then EPO 12,000 IU, IV, on Day 7, 8, and 9 of study participation
  Interventions: Drug: human chorionic gonadotropin (hCG), then epoetin alfa (EPO)
- NTx®-265 High Dose (Experimental): hCG 385 µg (10,000 IU), SC, on Day 1, 3 and 5 of study participation, then EPO 20,000 IU, IV, on Day 7, 8, and 9 of study participation
  Interventions: Drug: human chorionic gonadotropin (hCG), then epoetin alfa (EPO)
- Saline Placebo (Placebo Comparator)
  Interventions: Drug: Saline Placebo

INTERVENTIONS:
Drug: human chorionic gonadotropin (hCG), then epoetin alfa (EPO) — hCG 385 µg (10,000 IU), SC, on Day 1, 3 and 5 of study participation, then EPO 4,000 IU, IV, on Day 7, 8, and 9 of study participation
  Other Names: Ovidrel; Ovitrelle; Epogen; Eprex
  Arms: NTx®-265 Low Dose
Drug: human chorionic gonadotropin (hCG), then epoetin alfa (EPO) — hCG 385 µg (10,000 IU), SC, on Day 1, 3 and 5 of study participation, then EPO 12,000 IU, IV, on Day 7, 8, and 9 of study participation
  Other Names: Ovidrel; Ovitrelle; Epogen; Eprex
  Arms: NTx®-265 Medium Dose
Drug: human chorionic gonadotropin (hCG), then epoetin alfa (EPO) — hCG 385 µg (10,000 IU), SC, on Day 1, 3 and 5 of study participation, then EPO 20,000 IU, IV, on Day 7, 8, and 9 of study participation
  Other Names: Ovidrel; Ovitrelle; Epogen; Eprex
  Arms: NTx®-265 High Dose
Drug: Saline Placebo — Saline SC, on Day 1, 3, and 5 of study participation, then Saline IV, on Day 7, 8, and 9 of study participation
  Other Names: Sodium Chloride 0.9%
  Arms: Saline Placebo

SUMMARY:
The purpose of this study is:

* To assess the neurological outcome in acute ischemic stroke patients treated with NTx®-265, when compared with patients given a placebo control.
* To assess the safety and tolerability of NTx®-265 when given to acute ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* NIHSS score 8-20
* Stroke is ischemic in origin, supratentorial, and radiologically confirmed
* Patient is 24-48 hours from time of stroke onset when the first dose of NTx®-265 therapy is administered
* Reasonable expectation of availability to receive the full 9 day NTx®- 265 therapy and subsequent follow-up visits
* Reasonable expectation that patient will receive standard post-stroke physical, occupational, speech, and cognitive therapy as indicated
* Female patient is either not of childbearing potential or agrees to use two of the effective separate non-hormonal forms of contraception throughout the study

Exclusion Criteria:

* Patients presenting with lacunar, hemorrhagic and/or brain stem stroke
* Patients who have received tissue plasminogen activator (tPA)following the index stroke
* Patients classified as comatose
* Women who have tested positive for pregnancy, or are breast-feeding, or are not using a birth control
* Serum hemoglobin > 16 grams(g)/deciliter (dL)(males) or > 14 g/dL (females); or platelet count > 400,000/cubic millimeters(mm3)
* Advanced liver, kidney, cardiac, or pulmonary disease
* Elevated serum bilirubin,alkaline phosphatase, aspartate aminotransferase (AST) or alanine transaminase (ALT),creatinine, or prostate-specific antigen (PSA) levels
* Patients with a known history of hypercoagulability
* Expected survival < 1 year
* Allergy or other contraindication to hCG or EPO
* A known diagnosis of cancer in the previous 5 years
* Uncontrolled hypertension
* Use of either hCG or epoetin alfa within the previous 90 days
* Any condition known to elevate hCG
* Patients with a pre-stroke/pre-morbid modified Rankin Score (mRS)≥ 2
* Any patients not living independently
* Any other medical condition or degree of stroke such that, in the investigator's opinion, the patient should not be included in the trial
* With the exception of the qualifying stroke, any other stroke within the previous 3 months
* Patients who cannot take anti-platelet or anti-coagulant therapy
* Pre-existing and active major psychiatric or other chronic neurological disease
* Alcohol abuse or have a history of substance abuse or dependency within 12 months prior to the study
* Currently participating in another investigational study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Cramer, MD, Principal Investigator — Department of Neurology, University of California, Irvine Medical Center; Michael D Hill, MD, Principal Investigator — Department of Clinical Neurosciences, University of Calgary
Locations (23):
- University of California, Irvine Medical Center, Orange, California, United States
- Canada (4):
  - Foothills Medical Center , University of Calgary, Calgary, Alberta
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Neurological Institute, Montreal, Quebec
- India (18):
  - Lalitha Super Specialty Hospitals Pvt.Ltd, Guntur, Andhra Pradesh
  - Care Hospital, Hyderabad, Andhra Pradesh
  - Krishna Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - St.Theresa's General Hospital, Hyderabad, Andhra Pradesh
  - Apollo Hospitals, Hyderabad, Andhra Pradesh
  - Owaisi Hospital and Research Centre, Hyderabad, Andhra Pradesh
  - Mediciti Hospital, Hyderabad, Andhra Pradesh
  - Kamineni Hospital, Hyderabad, Andhra Pradesh
  - DBR & SK Super Speciality Hospital, Tirupati, Andhra Pradesh
  - Latha Superspecialities Hospital, Vijayawada, Andhra Pradesh
  - Suraksha Neuro Centre, Vijayawada, Andhra Pradesh
  - M S Ramaiah Memorial Hospital, Bangalore, Karnataka
  - J.S.S Medical College & Hospital, Bangalore, Karnataka
  - Ananthapuri Hospitals and Research Institute, Thiruvananthapuram, Kerala
  - Max Super Speciality Hospital, New Delhi, National Capital Territory of Delhi
  - Christian Medical College and Hospital, Ludhiana, Punjab
  - Vijaya Health Center, Chennai, Tamil Nadu
  - Christian Medical College Hospital, Vellore, Tamil Nadu

REFERENCES:
- [Derived] Cramer SC, Hill MD; REGENESIS-LED Investigators. Human choriogonadotropin and epoetin alfa in acute ischemic stroke patients (REGENESIS-LED trial). Int J Stroke. 2014 Apr;9(3):321-7. doi: 10.1111/ijs.12260. Epub 2014 Mar 3. PMID 24588854

RESULTS

PARTICIPANT FLOW:
Groups:
- NTx®-265 Low Dose: human chorionic gonadotropin (hCG) 385 µg (10,000 international unit [IU]), subcutaneously (SC), on Day 1, 3 and 5 of study participation, then epoetin alfa (EPO) 4,000 IU, intravenously (IV), on Day 7, 8, and 9 of study participation
- Placebo: saline SC, on Day 1, 3 and 5 of study participation, then saline IV, on Day 7, 8, and 9 of study participation
Period: Cohort 1
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Placebo
Started | 24 | 0 | 0 | 8
Completed | 22 | 0 | 0 | 6
Not Completed | 2 | 0 | 0 | 2
Period: Cohort 2
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Placebo
Started | 0 | 24 | 0 | 8
Completed | 0 | 18 | 0 | 6
Not Completed | 0 | 6 | 0 | 2
Period: Cohort 3
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Placebo
Started | 0 | 0 | 24 | 8
Completed | 0 | 0 | 20 | 7
Not Completed | 0 | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- NTx®-265 Low Dose: hCG 385 µg (10,000 IU), SC, on Day 1, 3 and 5 of study participation, then EPO 4,000 IU, IV, on Day 7, 8, and 9 of study participation
- Saline Placebo: saline SC, on Day 1, 3 and 5 of study participation, then saline IV, on Day 7, 8, and 9 of study participation
- Total: Total of all reporting groups
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Saline Placebo | Total
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 17 | 17 | 12 | 67
  >=65 years | 3 | 7 | 7 | 12 | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 57.42 (10.49) | 58.58 (13.32) | 54.83 (12.98) | 61.67 (12.38) | 58.13 (12.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 17 | 16 | 65
  Male | 6 | 10 | 7 | 8 | 31
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 2 | 0 | 0 | 2
  India | 24 | 22 | 24 | 24 | 94

OUTCOME MEASURES:

1. Primary Outcome: National Institutes of Health Stroke Scale (NIHSS) Change From Baseline at Day 90
Description: The NIHSS is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. Values range from 0 (no deficit) to 42 (dead).
Time Frame: Baseline and Day 90
Population: The analysis was conducted using a modified Intent-to-Treat population, defined as all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Saline Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24
scores on a scale | 6.79 (4.22) | 6.50 (4.53) | 6.08 (3.30) | 7.17 (4.24)

2. Secondary Outcome: NIHSS Response >=4 at Day 90
Description: The NIHSS is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. Values range from 0 (no deficit) to 42 (dead). NIHSS Response >=4 is defined as a >=4 change from baseline at Day 90.
Time Frame: Baseline and Day 90
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Saline Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24
participants
  No Response (<4) | 6 | 7 | 5 | 5
  Response (>=4) | 18 | 17 | 19 | 19

3. Secondary Outcome: NIHSS Change From Baseline at Day 30
Description: as for outcome 1
Time Frame: Baseline and Day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Saline Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24
scores on a scale | 4.67 (4.53) | 4.29 (3.37) | 5.00 (2.98) | 5.33 (3.33)

4. Secondary Outcome: Modified Rankin Scale (mRS) Response <=2 at Day 90
Description: The mRS measures the degree of disability or dependence in the daily activities of people who have suffered a stroke. The scale runs from 0 (perfect health without symptoms) to 6 (dead). mRS response <=2 is defined as the mRS score <=2 at Day 90.
Time Frame: Day 90
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Saline Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24
participants
  response (mRS <=2) | 11 | 11 | 15 | 18
  No response (mRS > 2) | 13 | 13 | 9 | 6

5. Secondary Outcome: Barthel Index at Day 90
Description: The Barthel Index measures 10 activities of daily living and mobility. A score of 100 = is best (able to live at home with a degree of independence), 0 is worst.
Time Frame: Day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Saline Placebo
Number analyzed (Participants) | 22 | 18 | 20 | 19
Scores on a scale | 68.18 (29.62) | 80.17 (22.04) | 85.25 (20.28) | 90.89 (12.69)

6. Secondary Outcome: Action Research Arm Test (ARAT) Change From Baseline at Day 90
Description: The ARAT assesses recovery of arm function following stroke through a series of subtests judging ability to grasp, grip, pinch, or move the arm; scores are on a scale; The total maximum (best) score is 57 and the total minimum (worst) score is 0.
Time Frame: Baseline and Day 90
Population: Not all patients enrolled in the group completed this outcome measure.
  The analysis was conducted using a modified Intent-to-Treat population, defined as all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Saline Placebo
Number analyzed (Participants) | 6 | 6 | 3 | 4
scores on a scale | 10.67 (13.37) | 33.50 (26.12) | 30.33 (16.80) | 23.75 (20.27)

7. Secondary Outcome: Gait Velocity Test Change From Baseline at Day 90
Description: The Gait Velocity Test assesses ability to walk as measured by the time (seconds) it takes a patient to walk 10 meters.
Time Frame: Baseline and Day 90
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Saline Placebo
Number analyzed (Participants) | 4 | 3 | 5 | 5
seconds | -22.75 (41.60) | -50.33 (48.95) | -6.40 (7.37) | -53.80 (54.15)

8. Secondary Outcome: Boston Naming Test (BNT) Change From Baseline at Day 90
Description: The BNT assesses impairment of language ability by asking patients to identify 20 different pictures each time the test is taken. A score of 20 is best, 0 is worst.
Time Frame: Baseline and Day 90
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Saline Placebo
Number analyzed (Participants) | 14 | 12 | 10 | 13
Scores on a scale | 3.93 (3.10) | 4.17 (4.11) | 0.20 (2.74) | 3.69 (3.82)

9. Secondary Outcome: Line Cancellation Test Change From Baseline at Day 90
Description: The Line Cancellation Test detects the loss of awareness of one side of the body. A score of 0.00 (no units) is normal (patient favors neither right nor left side). A score of +1.00 indicates severe unawareness of the left side. A score of -1.00 indicates severe unawareness of the right side.
Time Frame: Baseline and Day 90
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Saline Placebo
Number analyzed (Participants) | 7 | 10 | 10 | 9
scores on a scale | -0.03 (0.03) | -0.07 (0.11) | -0.04 (0.10) | -0.00 (0.16)

10. Secondary Outcome: Trails A Test Change From Baseline at Day 90
Description: The Trails A test measures visual scanning, numeric sequencing, and visual-motor coordination; the test score is the time (seconds) required to connect 25 numbers (e.g., 1, 2, 3, 4…)
Time Frame: Baseline and Day 90
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Saline Placebo
Number analyzed (Participants) | 6 | 9 | 7 | 9
seconds | -11.33 (22.20) | -21.89 (22.10) | -13.29 (21.91) | -23.44 (25.53)

11. Secondary Outcome: Trails B Test Change From Baseline at Day 90
Description: The Trails B test measures visual scanning, numeric sequencing, and visual-motor coordination; the test score is the time (seconds) required to connect 25 alpha numeric circles (e.g., 1, A, 2, B, 3, C, 4, D)
Time Frame: Baseline and Day 90
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Saline Placebo
Number analyzed (Participants) | 6 | 6 | 7 | 9
seconds | -44.33 (51.60) | -41.33 (62.89) | -55.14 (59.92) | -22.78 (71.22)

12. Secondary Outcome: Geriatric Depression Scale at Day 90
Description: The Geriatric Depression Scale is commonly used to assess depression in stroke patients of any age by asking 15 yes/no questions, and then scored. A score of 0 - 5 is normal, whereas a score of 6 -15 suggests depression.
Time Frame: Day 90
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Saline Placebo
Number analyzed (Participants) | 20 | 17 | 18 | 19
scores on a scale | 7.25 (4.24) | 3.88 (3.08) | 3.56 (2.77) | 4.74 (3.90)

ADVERSE EVENTS:
Time Frame: Adverse events were captured from the time of first dose to Day 30. Serious adverse events were captured from the time of first dose to Day 90.
Arm/Group | NTx®-265 Low Dose | NTx®-265 Medium Dose | NTx®-265 High Dose | Saline Placebo
Serious Adverse Events (participants affected / at risk) | 2/24 | 4/24 | 3/24 | 2/24
Other Adverse Events (participants affected / at risk) | 9/24 | 19/24 | 2/24 | 10/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NTx®-265 Low Dose (N=24) | NTx®-265 Medium Dose (N=24) | NTx®-265 High Dose (N=24) | Saline Placebo (N=24)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Cerebral Vascular Accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhagic Transformation Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischemic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden Cardiac Death (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ventricular Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NTx®-265 Low Dose (N=24) | NTx®-265 Medium Dose (N=24) | NTx®-265 High Dose (N=24) | Saline Placebo (N=24)
Depression (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 6 (6) | 0 (0) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomitting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was terminated after 96 of a planned 128 patients were enrolled, thus limiting opportunities to demonstrate a clear statistical benefit of active therapy compared to placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days